CLINICAL TRIAL: NCT06736405
Title: Effect of Pericapsular Nerve Group Block on Postoperative Cognitive Function in Total Hip Replacement Surgery
Brief Title: Effect of Pericapsular Nerve Group Block on Postoperative Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: POCD
Record Dates: First submitted 2024-11-13; First posted 2024-12-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Total Hip Replacement; Pericapsular Nerve Group Bloc; Postoperative Cognitive Dysfunction
Keywords: Total hip replacement; Pericapsular nerve group bloc; Postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group block (Active Comparator): Pericapsular nerve group block will be applied to patients in addition to standard treatment to prevent postoperative pain.
  Interventions: Other: Pericapsular nerve group block
- No Pericapsular nerve group block (Active Comparator): Pericapsular nerve group block will be applied to patients in addition to standard treatment to prevent postoperative pain.
  Interventions: Other: No Pericapsular nerve group block

INTERVENTIONS:
Other: Pericapsular nerve group block — Pericapsular nerve group block will be applied to patients in addition to standard treatment to prevent postoperative pain
  Arms: Pericapsular nerve group block
Other: No Pericapsular nerve group block — Patients will be given standard treatment to prevent postoperative pain
  Arms: No Pericapsular nerve group block

SUMMARY:
The aim of this study was to examine the effect of pericapsular nerve group (PENG) block, which is frequently applied for postoperative analgesia in total hip replacement surgeries performed under spinal anesthesia, on postoperative cognitive function in patients aged 65 years and older.

The main question of the study is as follows:

Can the analgesic effect of preoperative PENG block without causing motor block in total hip replacement surgeries performed under spinal anesthesia in patients aged 65 years and older reduce the incidence of postoperative cognitive dysfunction (POCD)?

DETAILED DESCRIPTION:
Patients aged 65 years and older, with (American Society of Anesthesiologists) ASA physical status I, II and III, and scheduled for total hip arthroplasty surgery under spinal anesthesia will be included in the study. Patient characteristics (age, gender, body mass index, etc.), Confusion Assessment Method (CAM), Yesavage Geriatric Depression Scale, Frail Frailty and Mini-Mental State Examination (MMSE) performed face-to-face will be recorded. Preoperatively, 24-72 hours before, patients' cognitive functions will be re-evaluated out of 26 points with telephone versions of the MMSE (T-MMSE). Intraoperatively, surgical duration, dermatomal block level due to spinal anesthesia, ephedrine or atropine requirement, pulse and blood pressure values will be recorded during the surgery. One group will receive a single dose ipsilateral pericapsular nerve group (PENG) block (20 ml 0.25% plain bupivacaine) under ultrasound guidance before surgery. The other group will receive a sham block. Cognitive function of the patients will be evaluated with T-MMSE on the 1st, 7th, 30th and 90th days postoperatively. Postoperative pain status of the patients will be recorded face-to-face at 0, 2, 8, 16, 24 and 48 hours, and via telephone on the 7th, 30th and 90th days with numerical rating scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo surgery with spinal anesthesia due to total hip replacement
* ASA (American Society of Anesthesiologists) I-II-III patients
* Patients aged 65 and over
* Patients with a preoperative fasting period of approximately 8 hours

Exclusion Criteria:

* Refusal to participate in the study
* ASA (American Society of Anesthesiologists) score of 4 and above
* Body mass index >40 kg/m²)
* Failure of spinal block
* Patients who underwent surgery with general anesthesia
* Patients who received preoperative and intraoperative sedation
* Patients who will undergo revision surgery
* Patients with a history of drug use
* Patients with psychiatric disorders or those taking antipsychotic medications (depression, bipolar disorder, schizophrenia, etc.)
* Patients with central nervous system disease (Alzheimer's disease, Parkinson's disease, multiple sclerosis, etc.)
* Patients who do not accept spinal anesthesia and/or pericapsular nerve group (PENG) block
* Patients with a preoperative Mini Mental Test (MMT) score below 25
* Patients with contraindications for regional anesthesia techniques
* Patients who developed perioperative delirium
* Patients with visual or hearing impairment
* Patients who require blood or blood product transfusion during surgery
* Patients who cannot cooperate in the postoperative period

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Frequency of postoperative cognitive dysfunction (POCD) | 3 months
  The primary outcome of the study was the frequency of postoperative cognitive dysfunction (POCD). Postoperative cognitive function of the patients will be evaluated with telephone versions of the Mini-Mental State Examination (T-MMSE) between 0 and 26 points. Higher scores indicate better cognitive function. POCD was defined as a decline of ≥1 standard deviation (SD) from the baseline T-MMSE score, observed at postoperative day 7, day 30, or day 90.

SECONDARY OUTCOMES:
11 - point numerical rating scale (NRS) | 3 months
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained
Mobilization | 3 days
  The time from the patient's first assisted mobilization start will be recorded in hours
Rescue analgesic requirement | 3 days
  Number of additional analgesic applications
Discharge time | 7 days
  Postoperative hospital discharge time

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No